CLINICAL TRIAL: NCT07332351
Title: Intravesical Nadofaragene Firadenovec With Neoadjuvant Chemotherapy and Durvalumab in Patients With Muscle Invasive Bladder Cancer (TRIFECTA)
Brief Title: Neoadjuvant Intravesical Nadofaragene Firadenovec With Gemcitabine, Cisplatin and Durvalumab for the Treatment of Muscle Invasive Bladder Cancer, TRIFECTA Trial
Acronym: TRIFECTA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1126027; NCI-2025-09407 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2026-01-06; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma; Stage II Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8
Keywords: Urinary Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Synapsins; durvalumab; Immunoglobulin G; Disulfides; Gemcitabine; Cisplatin; Cystectomy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (durvalumab, chemotherapy, nadofaragene firadenovec) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1, gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV on day 1 or days 1 and 8 of each cycle. Patients also receive nadofaragene firadenovec intravesically on day 1 of cycles 1 and 4. Cycles repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Starting 4-8 weeks after treatment, patients undergo RC per standard clinical care. Following RC, patients may receive durvalumab at the discretion of the clinician. Additionally, patients undergo urine and blood sample collection and CT, MRI or PET/CT throughout the study.
  Interventions: Biological: Nadofaragene Firadenovec; Biological: Durvalumab; Drug: Gemcitabine; Drug: Cisplatin; Procedure: Radical Cystectomy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Biological: Nadofaragene Firadenovec — Given intravesically
  Other Names: Adstiladrin; Instiladrin; Recombinant Adenovirus-Interferon SCH 721015; Recombinant Adenovirus-Interferon With Syn3; Recombinant Adenovirus-Interferon/Syn3; SCH 721015
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1; Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain); Disulfide with Human Monoclonal MEDI4736 Kappa-chain; MEDI 4736
Drug: Gemcitabine — Given IV
Drug: Cisplatin — Given IV
  Other Names: Cisplatinum; Platinol
Procedure: Radical Cystectomy — Undergo RC
  Other Names: RC
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CT; CT Scan; CAT Scan
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: PET; PET Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI

SUMMARY:
This phase II trial tests the effect of intravesical nadofaragene firadenovec in combination with gemcitabine, cisplatin and durvalumab before (neoadjuvant) radical cystectomy (RC) in treating patients with muscle invasive bladder cancer. The combination of gemcitabine, cisplatin and durvalumab are already considered standard of care in the treatment of muscle invasive bladder cancer. This trial attempts to determine whether the addition of nadofaragene firadenovec to the current standard regiment is safe and can improve oncological outcomes for those with muscle invasive bladder cancer.

Nadofaragene firadenovec, a type of intravesical gene therapy, is a weakened adenovirus that carries a copy of the gene for interferon alfa-2b. This medication gets absorbed by the bladder and stimulates the bladder to naturally create interferon alfa-2b, which is thought to kill bladder cancer. Nadofaragene firadenovec is given in a solution that is placed directly into the bladder (intravesical) using a thin tube called a catheter. It is a medication that is already FDA approved for the treatment of non-muscle invasive bladder cancer. Gemcitabine is a chemotherapy drug that blocks the cells from making deoxyribonucleic acid and may kill tumor cells. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive standard of care neoadjuvant therapies for muscle invasive bladder cancer including: durvalumab intravenously (IV) over 60 minutes on day 1, gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV on day 1 or days 1 and 8 of each cycle. In addition, patients also receive nadofaragene firadenovec intravesically on day 1 of cycles 1 and 4. Cycles repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Starting 4-8 weeks after treatment, patients undergo RC per standard clinical care. Following RC, patients may receive durvalumab at the discretion of the clinician. Additionally, patients undergo urine and blood sample collection and computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET)/CT throughout the study.

After completion of study treatment, patients are followed for up to 30 days post-cystectomy to monitor for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of screening
* Ability to understand and willingness to sign the written informed consent document
* Patients with confirmed muscle-invasive urothelial carcinoma of the bladder (cT2-4a, N0-1, M0 or cT1, N1, M0), who are planning to undergo RC
* Pure urothelial or mixed histologic subtypes are allowed if urothelial is the primary histology (regardless of the % of conventional urothelial histology)
* Eligible to receive neoadjuvant cisplatin/gemcitabine and durvalumab per the patient's medical oncologist's discretion
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Hemoglobin count ≥ 9 gm/dL
* Absolute neutrophil count of ≥ 1500 cells/uL
* Platelet count of ≥ 100,000/uL
* Alanine and aspartate aminotransferase levels ≤ 2.5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN (≤ 2.5 x ULN for Gilbert syndrome)
* Creatinine clearance or estimated glomerular filtration rate (GFR) ≥ 40ml/min (using Chronic Kidney Disease Epidemiology Collaboration Formula [CKD-EPI] 2021 equation)
* For patients with evidence of, or history of HIV, chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, the viral load must be undetectable, or the infection must have been treated and cured. Patients are not allowed to be on immunosuppressive agents for HIV, HBV or HCV. Routine testing for HIV, HBV and HCV is not required for patients without such history unless clinically indicated
* Individuals with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are allowed to enroll

Exclusion Criteria:

* cT4b, N2-3, or M1 stage at time of screening
* Any known concurrent clinically relevant malignancies
* Prior systemic therapy for muscle-invasive bladder carcinoma (MIBC) (prior intravenous pembrolizumab for non-muscle invasive bladder carcinoma [NMIBC] is allowed)
* Current or prior use of systemic immunosuppressive medication within 14 days before first dose of investigational product. The following are allowed (not systemic route): intranasal, inhaled, intra-articular, topical steroids, local steroid injections
* Pure non-urothelial histology subtype/variant or any neuroendocrine (small or large cell) component
* Prior treatment with adenovirus-based drugs
* Known hypersensitivity or allergy to any components of rAd-interferon (IFN)a/Syn3
* Currently receiving other investigational agent
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) on radical cystectomy (RC) specimen | At time of radical cystectomy (RC), approximately 4-8 weeks following completion of neoadjuvant systemic therapies
  Will be defined as the proportion of participants achieving ypT0N0. Will employ Simon's optimal two-stage design (Simon, 1989) to test the null hypothesis that the true pCR rate is 33.8% versus the alternative hypothesis of 56%. The observed pCR rate will be reported with an exact 95% confidence interval using the Clopper-Pearson method.
Downstaging (≤ ypT1N0) on RC specimen | At time of radical cystectomy (RC), approximately 4-8 weeks following completion of neoadjuvant systemic therapies

SECONDARY OUTCOMES:
Proportion of patients who undergo RC | Within 10 weeks from last neoadjuvant therapy dose
  Will be defined as the number of patients who ultimately receive RC divided by the total number of patients that receive at least one administration of neoadjuvant therapy.
Incidence of grade 3 or higher treatment-related adverse events (AE) | From initiation of neoadjuvant systemic therapies (day 1 of cycle 1; 4 cycles total; each cycle is 21 days), through 30 days post-RC (RC occurs approximately 4-8 weeks after completion of neoadjuvant systemic therapies)
  Will be graded by provider-scored toxicity via the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will be summarized descriptively, including the number and proportion of patients experiencing at least one grade ≥ 3 AE, and the type, severity, and relatedness of all treatment-related AEs, attributed by agent.
Incidence of AEs | From initiation of neoadjuvant systemic therapies (day 1 of cycle 1; 4 cycles total; each cycle is 21 days), through 30 days post-RC (RC occurs approximately 4-8 weeks after completion of neoadjuvant systemic therapies)
  Will be summarized by maximum CTCAE grade and relatedness to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wright, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No